CLINICAL TRIAL: NCT04659031
Title: A Phase 1, Open-Label, Single and Multiple Ascending Dose Study of ABC008 in Adult Patients With Inclusion Body Myositis (IBM)
Brief Title: A Phase 1 Study of ABC008 in Ascending (Single Ascending Dose/Multiple Ascending Dose) Study in Patients With (IBM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abcuro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABC008-IBM-101
Record Dates: First submitted 2020-11-25; First posted 2020-12-09 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-06

CONDITIONS: Inclusion Body Myositis
Keywords: Inclusion Body Myositis; IBM
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Cohort D1 (Experimental): Single Dose 0.1 mg / kg ABC008
  Interventions: Drug: ABC008
- Cohort D2 (Experimental): Single Dose 0.5 mg / kg ABC008
  Interventions: Drug: ABC008
- Cohort D3 (Experimental): Single Dose 2.0 mg / kg ABC008
  Interventions: Drug: ABC008
- Cohort D4 (Experimental): Single Dose 5.0 mg / kg ABC008
  Interventions: Drug: ABC008
- Cohort D5 (Experimental): X.X mg / kg ABC008
  Interventions: Drug: ABC008
- Cohort 6 (Experimental): Single 2.0 mg / kg ABC008
  Interventions: Drug: ABC008
- MAD Phase Cohort 1 (Experimental): Multiple Dose 0.1 mg / kg ABC008 every 8 weeks
  Interventions: Drug: ABC008
- MAD Phase Cohort 2 (Experimental): Multiple Dose 0.5 mg / kg ABC008 every 8 weeks
  Interventions: Drug: ABC008
- MAD Phase Cohort 3 (Experimental): Multiple Dose 2.0 mg / kg ABC008 every 8 weeks
  Interventions: Drug: ABC008

INTERVENTIONS:
Drug: ABC008 — ABC008

SUMMARY:
An open-label, ascending dose study for adult patients with Inclusion Body Myositis (IBM).

DETAILED DESCRIPTION:
Participants who successfully complete the SAD EOT visit, and have no emerging safety issues, will be eligible to enroll in Part 2 (MAD). Eligible participants for the MAD part will have inclusion and exclusion criteria (same as those for Part 1) reviewed prior to dosing on MAD Day 1.

Participants who successfully complete the MAD EOT visit, and have no emerging safety issues, will be eligible to enrol in Part 3, MAD Extension.

After the final MAD visit (W48), participants will have the option to continue on to Part 3 MAD Extension.

For Part 3 (MAD Extension), participant dosing will be at 8-week intervals starting at Day 1. Duration of dosing in Part 3 will be up to approximately 80 weeks (18 months), or until a new long-term extension study has been initiated. The SMC will review all participant safety data approximately every 6 months while the Part 3 dosing continues.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of either clinico-pathologically defined IBM, clinically defined IBM, or probable IBM according to the European Neuromuscular Center (ENMC) IBM 2011
* Able to arise from a chair (with or without armrests) without support from another person or device
* Able to ambulate at least 20 feet / 6 meters with or without assistive device

Exclusion Criteria:

* Taking > 7.5 mg prednisolone (or equivalent) or on intravenous immunoglobulin (IVIg) or other immunosuppressants within the last 3 months. Topical, nasal, and ocular corticosteroids are allowed unless they are being widely applied or the severity of the underlying condition makes them unsuitable in the Investigator's opinion. Local steroid injections are allowed

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety and Tolerability | Through Study Completion an average of 28 weeks for SAD (Single Ascending Dose) phase and 52 weeks for MAD (Multiple Ascending Dose) phase]
  Characterize the safety and tolerability profile of single (SAD) and multiple (MAD) escalating dose levels of ABC008 in IBM when administered subcutaneously (SC) as measured by the number and severity of treatment emergent adverse events, serious adverse events, and adverse events of special interest, number of dose limiting toxicities.

SECONDARY OUTCOMES:
Assessment of peak serum concentration (Cmax) | Day 1 and throughout the 24 weeks of follow up
  Assess the peak serum concentration (Cmax) of a single dose of ABC008
Assessment of time to peak serum concentration (Tmax) | Day 1 and throughout the 24 weeks of follow up
  Assess the time to peak serum concentration (Tmax) of a single dose of ABC008
Assessment of terminal half-life (t½) | Day 1
  Assess the terminal half-life (t½) of ABC008
Assessment of area under the concentration versus time curve from time zero to 24 hours post-dose (AUC0-24hr) | Day 1
  Assess the area under the concentration versus time curve of a single dose of ABC008 from time zero to 24 hours post-dose (AUC0-24hr)
Assessment of apparent clearance (CL/F) | Day 1 and throughout the 24 weeks of follow up
  Assessment of apparent clearance (CL/F) of a single dose of ABC008
Assessment of apparent volume of distribution (Vz/F) | Day 1 and throughout the 24 weeks of follow up
  Assessment of apparent volume of distribution (Vz/F) of a single dose of ABC008
Characterization of changes in KLRG1 expressing lymphocytes | Day 1 and throughout the 24 weeks of follow up
  Characterize changes in KLRG1 expressing lymphocytes
Qualitative assessment of [ 89Zr]Zr-Df-crefmirlimab | [Through Study Completion, avg. 48 weeks
  Qualitative assessment of [ 89Zr]Zr-Df-crefmirlimab uptake in involved skeletal muscles including inflamed and non-inflamed sites as determined by using a visual scoring (VS) system for the time point assessed, the possible scores VS1-VS5
Assessment of global distribution of [ 89Zr]Zr-Df-crefmirlimab uptake in skeletal muscle | [Through Study Completion, avg. 48 weeks
  Assessment of global distribution of [ 89Zr]Zr-Df-crefmirlimab uptake in skeletal muscle; Pattern(s) of absolute and relative changes in uptake within various skeletal muscle groups; Homogenous/diffuse, Focal, Mixed, Other
Assessment of global distribution of [ 89Zr]Zr-Df-crefmirlimab uptake in lymphoid organs | [Through Study Completion, avg. 48 weeks
  Assessment of global distribution of [ 89Zr]Zr-Df-crefmirlimab uptake in lymphoid organs; Uptake and relative changes in uptake within lymphoid tissue including spleen and lymph nodes as well as other T-cell rich tissues such as bone marrow
Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab pre and post dosing of ABC008 | [Through Study Completion, avg. 48 weeks
  Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab uptake and relative changes in uptake within inflamed muscle tissue through Positron Emission Tomography (PET)/computed tomography (CT) imaging pre- and post-dosing with ABC008
Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab, determined by standardized uptake value (SUV)-based quantitative analysis peak (SUVpeak) | [Through Study Completion, avg. 48 weeks
  Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab uptake in involved skeletal muscles including inflamed and non-inflamed sites, and measurement of magnitude of difference observations as determined by standardized uptake value (SUV)-based quantitative analysis peak (SUVpeak)
Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab, determined by standardized uptake value (SUV)-based quantitative analysis mean (SUVmean) | [Through Study Completion, avg. 48 weeks
  Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab uptake in involved skeletal muscles including inflamed and non-inflamed sites, and measurement of magnitude of difference observations as determined by standardized uptake value (SUV)-based quantitative analysis mean (SUVmean)
Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab, determined by standardized uptake value (SUV)-based quantitative analysis SUV of diseased muscle | [Through Study Completion, avg. 48 weeks
  Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab uptake in involved skeletal muscles including inflamed and non-inflamed sites, and measurement of magnitude of difference observations as determined by standardized uptake value (SUV)-based quantitative analysis SUV of diseased muscle
Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab, determined by standardized uptake value (SUV)-based quantitative analysis SUV reference tissue | [Through Study Completion, avg. 48 weeks
  Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab uptake in involved skeletal muscles including inflamed and non-inflamed sites, and measurement of magnitude of difference observations as determined by standardized uptake value (SUV)-based quantitative analysis SUV reference tissue
Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab, determined by standardized uptake value (SUV)-based quantitative analysis maximum (SUVmax) | [Through Study Completion, avg. 48 weeks
  Quantitative assessment of [ 89Zr]Zr-Df-crefmirlimab uptake in involved skeletal muscles including inflamed and non-inflamed sites, and measurement of magnitude of difference observations as determined by standardized uptake value (SUV)-based quantitative analysis maximum (SUVmax)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Brisbane, Herston
  - Perron Institute, Perth
  - Royal North Shore Hospital, Sydney

IPD SHARING:
Plan to Share IPD: Undecided